CLINICAL TRIAL: NCT02312960
Title: A Phase 4 Long-term Follow-up Study to Define the Safety Profile of Radium-223 Dichloride
Brief Title: Radium-223 Dichloride Long-term Follow-up Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16996; 2014-002407-25 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2025-01-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neoplasm Metastasis / Bone and Bones
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other): The subjects previously enrolled in a selected radium-223 dichloride feeder trial, their treating health care professional, or caregiver will be contacted in 6-month intervals for follow up and query.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — No study treatment will be provided in this long term follow up study.

SUMMARY:
Patients will be followed up in this study after prior treatment with BAY88-8223 / Radium-223 dichloride / Xofigo.

DETAILED DESCRIPTION:
This long-term follow up study will enroll subjects who will be transferred from selected interventional, company sponsored trials with radium-223 dichloride (feeder trials).

The primary objectives are to define the long term safety profile of radium-223 dichloride (for up to 7 years after the last dose of radium-223 dichloride); to assess the incidence of leukemia, myelodysplastic syndrome, aplastic anemia, and primary bone cancer or any other new primary malignancy; to assess the incidence of bone fractures and bone associated events (e.g., osteoporosis); and, in subjects who receive cytotoxic chemotherapy, to assess the incidence of febrile neutropenia and hemorrhage during their chemotherapy treatment and for up to 6 months thereafter at a frequency based on local clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously enrolled in a selected company sponsored feeder trial, and has received at least 1 dose of radium 223 dichloride or placebo in the feeder trial

Exclusion Criteria:

* Not applicable to this follow up study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (104):
- United States (15):
  - Anchorage, Alaska
  - Tucson, Arizona
  - Plantation, Florida
  - Indianapolis, Indiana
  - Ashland, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Omaha, Nebraska
  - Syracuse, New York
  - Pittsburgh, Pennsylvania
  - Watertown, South Dakota
  - Seattle, Washington
- Australia (4):
  - Darlinghurst, New South Wales
  - Westmead, New South Wales
  - Fitzroy, Victoria
  - Heidelberg, Victoria
- Belgium (2):
  - Kortrijk
  - Leuven
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - Barretos/SP, São Paulo
  - São Paulo, São Paulo
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Prague, Czechia
- Finland (2):
  - Helsinki
  - Tampere
- France (6):
  - Bordeaux
  - Nantes
  - Nîmes
  - Saint-Cloud
  - Tours
  - Villejuif
- Germany (11):
  - Ulm, Baden-Wurttemberg
  - Erlangen, Bavaria
  - München, Bavaria
  - Rostock, Mecklenburg-Vorpommern
  - Aachen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Magdeburg, Saxony-Anhalt
  - Jena, Thuringia
  - Berlin
  - Bremen
- Chai Wan, Hong Kong
- Israel (7):
  - Afula
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
  - Zrifin
- Italy (5):
  - Forlì Cesena, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Milan, Lombardy
  - Trento, Trentino-Alto Adige
- Japan (13):
  - Matsuyama, Ehime
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Kurashiki, Okayama-ken
  - Sayama, Osaka
  - Hidaka, Saitama
  - Kita-Adachigun, Saitama
  - Koto-ku, Tokyo
  - Fukuoka
  - Kumamoto
  - Miyazaki
  - Osaka
- Norway (2):
  - Bodø
  - Oslo
- Poland (3):
  - Bialystok
  - Gliwice
  - Warsaw
- Obninsk, Russia
- Singapore, Singapore
- South Korea (4):
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Incheon
  - Seoul
- Spain (8):
  - Badalona (Barcelona), Barcelona
  - Palma de Mallorca, Illes Baleares
  - A Coruña
  - Barcelona
  - Madrid
  - Málaga
  - Pamplona
  - Seville
- Umeå, Sweden
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- United Kingdom (8):
  - Truro, Cornwall
  - Plymouth, Devon
  - Sheffield, South Yorkshire
  - Guildford, Surrey
  - Sutton, Surrey
  - Coventry, Warwickshire
  - Bristol
  - Cottingham

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — https://www.clinicaltrialsregister.eu/ctr-search/search

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 22 countries between 18-Dec-2014 (first participant first visit) and 31-Jan-2024 (last participant last visit).
Pre-assignment Details: A total of 257 participants were screened from the selected feeder studies into the 16996 study for long-term follow-up. Of these, 255 participants entered the study and 2 participants did not complete screening.
Groups:
- From Study 15396 Radium-223 Dichloride+Abi/Pred Group: Safety follow up from feeder study 15396. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of National Institute of Standards and Technology [NIST] update) at intervals of every 4 weeks, along with abiraterone acetate plus prednisone/prednisolone (abi/pred) for up to 6 cycles.
- From Study 15396 Placebo+Abi/Pred Group: Safety follow up from feeder study 15396. Participants received placebo matched to radium-223 dichloride at intervals of every 4 weeks, along with abiraterone acetate plus prednisone/prednisolone (abi/pred) for up to 6 cycles.
- From Study 16216 Radium-223 Dichloride Group: Safety follow up from feeder study 16216. Participants received radium-223 dichloride 50 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group: Safety follow up from feeder study 16298. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks, along with single hormonal agent, for up to 6 cycles.
- From Study 16298 Placebo + Hormonal Therapy Group: Safety follow up from feeder study 16298. Participants received placebo matched to radium-223 dichloride at intervals of every 4 weeks, along with single hormonal agent for up to 6 cycles.
- From Study 16506 Radium-223 Dichloride Group: Safety follow up from feeder study 16506. Participants received radium-223 dichloride 50 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16507 Radium-223 Dichloride Treatment A Group: Safety follow up from feeder study 16507. Participants received radium-223 dichloride 55 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16507 Radium-223 Dichloride Treatment B Group: Safety follow up from feeder study 16507. Participants received radium-223 dichloride 88 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16507 Radium-223 Dichloride Treatment C Group: Safety follow up from feeder study 16507. Participants received radium-223 dichloride 55 kBg/kg at intervals of every 4 weeks for up to 12 cycles.
- From Study 16544 Radium-223 Dichloride+Abi/Pred Group: Safety follow up from feeder study 16544. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks, along with Abi/Pred for up to 6 cycles.
- From Study 16544 Radium-223 Dichloride+Enzalutamide Group: Safety follow up from feeder study 16544. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks, along with enzalutamide for up to 6 cycles.
- From Study 16544 Radium-223 Dichloride Group: Safety follow up from feeder study 16544. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks for up to 6 cycles.
- From Study 17096 Radium-223 Dichloride + EXE/EVE Group: Safety follow up from feeder study 17096. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) along with exemestane (EXE) + everolimus (EVE) once daily.
- From Study 17096 Placebo + EXE/EVEgroup: Safety follow up from feeder study 17096. Participants received placebo matched to radium-223 dichloride along with exemestane (EXE) + everolimus (EVE) once daily.
Period: Overall Study
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Started | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Completed | 14 | 15 | 3 | 3 | 3 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 5 | 9
Not Completed | 25 | 34 | 28 | 11 | 6 | 5 | 10 | 8 | 9 | 7 | 3 | 1 | 28 | 19
Not completed — Death | 24 | 32 | 25 | 11 | 5 | 5 | 8 | 5 | 7 | 3 | 3 | 1 | 25 | 19
Not completed — Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set during long-term follow up (SAF-LTF): All participants who have received at least 1 dose of radium-223 dichloride or placebo in an eligible feeder study and who have signed informed consent to 16996.
Groups:
- Total: Total of all reporting groups
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup | Total
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 3 | 9 | 5 | 2 | 1 | 2 | 5 | 1 | 1 | 1 | 26 | 16 | 81
  >=65 years | 33 | 46 | 28 | 5 | 4 | 3 | 10 | 7 | 6 | 8 | 3 | 2 | 7 | 12 | 174
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 14 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 28 | 84
  Male | 39 | 49 | 31 | 0 | 0 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 0 | 0 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 13
  Not Hispanic or Latino | 32 | 41 | 31 | 13 | 9 | 5 | 11 | 9 | 10 | 8 | 3 | 3 | 30 | 27 | 232
  Unknown or Not Reported | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 13 | 0 | 4 | 2 | 0 | 4 | 5 | 2 | 0 | 0 | 0 | 10 | 7 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 4
  White | 29 | 30 | 31 | 9 | 7 | 5 | 7 | 4 | 7 | 7 | 3 | 3 | 21 | 20 | 183
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radium-223 Dichloride-/Placebo-related Adverse Events (AEs)
Description: Adverse events considered related to radium-223 dichloride or placebo (received in the feeder studies), first arising or worsening on or after the date the participant signed the 16996 informed consent.
Time Frame: Up to 7 years
Population: SAF-LTF
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 3 | 0

2. Primary Outcome: Severity of Radium-223 Dichloride-/Placebo-related Adverse Events (AEs)
Description: Severity will be measured as per guidelines by Common Terminology Criteria for Adverse Events; Version 4.03 (CTCAE)
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants
  Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
  Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 (death) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Radium-223 Dichloride-/Placebo-related Serious Adverse Events
Description: Serious adverse events considered related to radium-223 dichloride or placebo (received in the feeder studies), first arising or worsening on or after the date the participant signed the 16996 informed consent.
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Leukemia
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Myelodysplastic Syndrome
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Aplastic Anemia
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Primary Bone Cancer
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Any Other New Primary Malignancy
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Bone Fractures
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 3 | 6 | 1 | 1 | 3 | 0 | 1 | 2 | 3 | 1 | 2 | 0 | 6 | 7

10. Primary Outcome: Number of Participants With Bone-associated Events
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 4 | 2 | 0 | 1 | 3 | 0

11. Primary Outcome: Number of Participants With Febrile Neutropenia in Subjects Who Receive Cytotoxic Chemotherapy
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0

12. Primary Outcome: Number of Participants With Hemorrhage in Subjects Who Receive Cytotoxic Chemotherapy
Time Frame: Up to 7 years
Measure: Number; unit: Participants
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
Number analyzed (Participants) | 39 | 49 | 31 | 14 | 9 | 5 | 11 | 9 | 11 | 9 | 4 | 3 | 33 | 28
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 7 years
Groups:
- From Study 15396 Radium-223 Dichloride+Abi/Pred Group: Safety FU from feeder study 15396. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of National Institute of Standards and Technology [NIST] update) at intervals of every 4 weeks, along with abiraterone acetate plus prednisone/prednisolone (abi/pred) for up to 6 cycles.
- From Study 15396 Placebo+Abi/Pred Group: Safety FU from feeder study 15396. Participants received placebo matched to radium-223 dichloride at intervals of every 4 weeks, along with abiraterone acetate plus prednisone/prednisolone (abi/pred) for up to 6 cycles.
- From Study 16216 Radium-223 Dichloride Group: Safety FU from feeder study 16216. Participants received radium-223 dichloride 50 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group: Safety FU from feeder study 16298. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks, along with single hormonal agent, for up to 6 cycles.
- From Study 16298 Placebo + Hormonal Therapy Group: Safety FU from feeder study 16298. Participants received placebo matched to radium-223 dichloride at intervals of every 4 weeks, along with single hormonal agent for up to 6 cycles.
- From Study 16506 Radium-223 Dichloride Group: Safety FU from feeder study 16506. Participants received radium-223 dichloride 50 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16507 Radium-223 Dichloride Treatment A Group: Safety FU from feeder study 16507. Participants received radium-223 dichloride 55 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16507 Radium-223 Dichloride Treatment B Group: Safety FU from feeder study 16507. Participants received radium-223 dichloride 88 kBg/kg at intervals of every 4 weeks for up to 6 cycles.
- From Study 16544 Radium-223 Dichloride+Abi/Pred Group: Safety FU from feeder study 16544. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks, along with Abi/Pred for up to 6 cycles.
- From Study 16544 Radium-223 Dichloride+Enzalutamide Group: Safety FU from feeder study 16544. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks, along with enzalutamide for up to 6 cycles.
- From Study 16544 Radium-223 Dichloride Group: Safety FU from feeder study 16544. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) at intervals of every 4 weeks for up to 6 cycles.
- From Study 17096 Radium-223 Dichloride + EXE/EVE Group: Safety FU from feeder study 17096. Participants received radium-223 dichloride 50 kBg/kg (55 kBq/kg after implementation of NIST update) along with exemestane (EXE) + everolimus (EVE) once daily.
- From Study 17096 Placebo + EXE/EVEgroup: Safety FU from feeder study 17096. Participants received placebo matched to radium-223 dichloride along with exemestane (EXE) + everolimus (EVE) once daily.
Arm/Group | From Study 15396 Radium-223 Dichloride+Abi/Pred Group | From Study 15396 Placebo+Abi/Pred Group | From Study 16216 Radium-223 Dichloride Group | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group | From Study 16298 Placebo + Hormonal Therapy Group | From Study 16506 Radium-223 Dichloride Group | From Study 16507 Radium-223 Dichloride Treatment A Group | From Study 16507 Radium-223 Dichloride Treatment B Group | From Study 16507 Radium-223 Dichloride Treatment C Group | From Study 16544 Radium-223 Dichloride+Abi/Pred Group | From Study 16544 Radium-223 Dichloride+Enzalutamide Group | From Study 16544 Radium-223 Dichloride Group | From Study 17096 Radium-223 Dichloride + EXE/EVE Group | From Study 17096 Placebo + EXE/EVEgroup
All-Cause Mortality (participants affected / at risk) | 24/39 | 32/49 | 25/31 | 11/14 | 5/9 | 5/5 | 8/11 | 5/9 | 7/11 | 3/9 | 3/4 | 1/3 | 25/33 | 19/28
Serious Adverse Events (participants affected / at risk) | 3/39 | 4/49 | 4/31 | 1/14 | 1/9 | 0/5 | 2/11 | 3/9 | 3/11 | 0/9 | 1/4 | 0/3 | 4/33 | 6/28
Other Adverse Events (participants affected / at risk) | 2/39 | 6/49 | 0/31 | 3/14 | 3/9 | 0/5 | 1/11 | 1/9 | 3/11 | 3/9 | 1/4 | 1/3 | 8/33 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | From Study 15396 Radium-223 Dichloride+Abi/Pred Group (N=39) | From Study 15396 Placebo+Abi/Pred Group (N=49) | From Study 16216 Radium-223 Dichloride Group (N=31) | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group (N=14) | From Study 16298 Placebo + Hormonal Therapy Group (N=9) | From Study 16506 Radium-223 Dichloride Group (N=5) | From Study 16507 Radium-223 Dichloride Treatment A Group (N=11) | From Study 16507 Radium-223 Dichloride Treatment B Group (N=9) | From Study 16507 Radium-223 Dichloride Treatment C Group (N=11) | From Study 16544 Radium-223 Dichloride+Abi/Pred Group (N=9) | From Study 16544 Radium-223 Dichloride+Enzalutamide Group (N=4) | From Study 16544 Radium-223 Dichloride Group (N=3) | From Study 17096 Radium-223 Dichloride + EXE/EVE Group (N=33) | From Study 17096 Placebo + EXE/EVEgroup (N=28)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | From Study 15396 Radium-223 Dichloride+Abi/Pred Group (N=39) | From Study 15396 Placebo+Abi/Pred Group (N=49) | From Study 16216 Radium-223 Dichloride Group (N=31) | From Study 16298 Radium-223 Dichloride+Hormonal Therapy Group (N=14) | From Study 16298 Placebo + Hormonal Therapy Group (N=9) | From Study 16506 Radium-223 Dichloride Group (N=5) | From Study 16507 Radium-223 Dichloride Treatment A Group (N=11) | From Study 16507 Radium-223 Dichloride Treatment B Group (N=9) | From Study 16507 Radium-223 Dichloride Treatment C Group (N=11) | From Study 16544 Radium-223 Dichloride+Abi/Pred Group (N=9) | From Study 16544 Radium-223 Dichloride+Enzalutamide Group (N=4) | From Study 16544 Radium-223 Dichloride Group (N=3) | From Study 17096 Radium-223 Dichloride + EXE/EVE Group (N=33) | From Study 17096 Placebo + EXE/EVEgroup (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (10) | 1 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device failure (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT02312960/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT02312960/SAP_001.pdf